CLINICAL TRIAL: NCT02381626
Title: DRIIVE (Data and Research on Interventions to Improve the Vehicular Environment)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York University (Other); New York State Department of Health (Other Government); The City College of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-247
Record Dates: First submitted 2015-02-24; First posted 2015-03-06 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-02

CONDITIONS: Vehicular Environment
Keywords: HEPA filter; 14-247
MeSH Terms: interventions — Surveys and Questionnaires

ARMS (2):
- Intervention Group (Experimental): During the first 2 weeks, measurements (e.g. biological markers and air monitoring) will be taken under usual conditions. At the end of the initial two weeks, portable HEPA air purifiers (136) will be placed in the Intervention Group drivers' cars and the air monitoring and biological parameters will be repeated for another 2-week period, to determine changes in PM levels and physiological measurements as a result of this targeted intervention.
  Interventions: Device: HEPA air purifier; Behavioral: questionnaires; Other: Log-book; Other: Urine sample
- Wait-list Control Group (Experimental): During the first 2 weeks, measurements (e.g. biological markers and air monitoring) will be taken under usual conditions. The Wait-list Control Group drivers will not receive a HEPA air purifier at this time, but will also have the air monitoring and biological parameters repeated for another 2 weeks. At the end of the 1 month period of measurements for both groups of drivers, the Wait-list drivers will then receive a HEPA air purifier, so that they may also potentially benefit from the intervention being tested in this study, but no further measurements will be taken.
  Interventions: Device: HEPA air purifier; Behavioral: questionnaires; Other: Log-book; Other: Urine sample

INTERVENTIONS:
Device: HEPA air purifier — air purifiers to remove PM and volatile organic compounds will be placed in drivers cars
Behavioral: questionnaires
Other: Log-book — PM and biological measurements
Other: Urine sample — PAH (Polycyclic Aromatic Hydrocarbon) will be assessed via urine sample collection of Urinary 1 hydroxy pyrene and particulate matter collected via Polyurethane Foam Filter (PUF) sampler

SUMMARY:
The purpose of this study is to look at air quality in cabs and see if the air quality inside taxi cabs is connected to increased risks for lung and heart health problems. Another purpose of the study is to see if putting an air filter inside the car may help improve the air quality and lower health risks.

This is important because air pollution can be harmful to health. Air pollution is made up of very tiny particles (things) floating in the air around us, called particulate matter. Particulate matter is made up of dust, smoke, dirt, and gas fumes and can get into our bodies as we breathe. It has been linked to risk for lung cancer and heart disease. It is important because taxi drivers spend many hours of their day inside their cars.

The investigators hope that this study will help them find out if using air filters inside cabs will help lower the levels of pollution in cabs and reduce its effects on the health of taxi drivers. They will use these results to educate the taxi driver community.

DETAILED DESCRIPTION:
DRIIVE (Data and Research on Interventions to Improve the Vehicular Environment) is a community-engaged translational pilot project that will utilize a three parallel arm design to obtain preliminary data on associations between Particulate Matter (PM)/air pollution and physiologic measurements and biomarkers in taxi drivers, and to determine the impact of a HEPA filter (to remove PM and volatile organic compounds) intervention on such physiologic measurements and biomarkers. DRIIVE is funded by the New York State Department of Health Empire Clinical Research Investigator Program (ECRIP), which trains physicians in clinical research in New York. Drivers will be randomized to one of two groups: Intervention or Wait-list Control. In total, two groups of 14 participants in each group will be recruited: 1) Wait List Control group, who will receive a HEPA filter at the end of the 1 month participation period, and 2) Intervention group, who will receive a HEPA filter two weeks into their participation period. The project will be completed within a 2 year timeframe.

ELIGIBILITY:
Inclusion Criteria:

Drivers:

* Full-time New York City cab drivers;
* Non Smokers (assessed by modified BRFSS smoking question within screening tool) ;
* Male;
* Between the ages of 21 and 90;
* No immediate plans (within the next 3 months) to leave the City for vacation or for trips back to their home country
* Driver for at least 3 years*;
* Driving schedule does not include overnight shifts, nor does driver have an additional job overnight;
* Own a smart phone (in order to collect heart rate variability data)
* Should self-report at least "Very well" level of English fluency (according to the standard US census question)
* Have working cigarette lighter receptacle/socket inside taxi cab *The requirement to have worked at least 3 years in the U.S. should minimize any acute health effects/disease due to high levels of contaminants associated with country of origin

Exclusion Criteria:

Drivers:

* Smoker or uses smokeless tobacco products;
* Resides in a smoking household (where 1 or more household members smoke);
* Has a sleep disorder (including insomnia, delayed sleep phase syndrome (DSPS), narcolepsy, night terror, sleep apnea, sleep walking);
* Has a current or previous diagnosis of any type of cancer;
* Has a diagnosis of an inflammatory, autoimmune, or chronic infectious disease (including rheumatoid arthritis, lupus, chronic liver disease, multiple sclerosis, fibromyalgia, inflammatory bowel disease, psoriasis, HIV);
* Has a serious cardiopulmonary medical condition (including cardiovascular disease, congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), restrictive lung disease, interstitial lung disease, asthma, acute or chronic bronchitis, cystic fibrosis, pneumonia, tuberculosis, pneumoconiosis, pulmonary hypertension, pulmonary embolism, pleural effusion, pneumothorax, obesity hypoventilation syndrome, neuromuscular lung disease).
* Self reports -well‖ level of English fluency and indicates a preference for an interpreter.

Ages: 21 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-12; Primary Completion 2020-10-18 (Actual); Study Completion 2020-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Leng, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: During the first 2 weeks, measurements (e.g. biological markers and air monitoring) will be taken under usual conditions. At the end of the initial two weeks, portable HEPA air purifiers (136) will be placed in the Intervention Group drivers' cars and the air monitoring and biological parameters will be repeated for another 2-week period, to determine changes in PM levels and physiological measurements as a result of this targeted intervention.
  HEPA air purifier: air purifiers to remove PM and volatile organic compounds will be placed in drivers cars
  questionnaires
  Log-book: PM and biological measurements
  Urine sample: PAH (Polycyclic Aromatic Hydrocarbon) will be assessed via urine sample collection of Urinary 1 hydroxy pyrene and particulate matter collected via Polyurethane Foam Filter (PUF) sampler
- Wait-list Control Group: During the first 2 weeks, measurements (e.g. biological markers and air monitoring) will be taken under usual conditions. The Wait-list Control Group drivers will not receive a HEPA air purifier at this time, but will also have the air monitoring and biological parameters repeated for another 2 weeks. At the end of the 1 month period of measurements for both groups of drivers, the Wait-list drivers will then receive a HEPA air purifier, so that they may also potentially benefit from the intervention being tested in this study, but no further measurements will be taken.
  HEPA air purifier: air purifiers to remove PM and volatile organic compounds will be placed in drivers cars
  questionnaires
  Log-book: PM and biological measurements
  Urine sample: PAH (Polycyclic Aromatic Hydrocarbon) will be assessed via urine sample collection of Urinary 1 hydroxy pyrene and particulate matter collected via Polyurethane Foam Filter (PUF) sampler
- Peer Non-driver: Peer non-driver (peer is matched to driver assigned to the HEPA filter intervention group)
Period: Overall Study
Arm/Group | Intervention Group | Wait-list Control Group | Peer Non-driver
Started | 17 | 16 | 6
Completed | 17 | 16 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Wait-list Control Group | Peer Non-driver | Total
Number analyzed (Participants) | 17 | 16 | 6 | 39
Age, Continuous [Mean (Full Range); unit: years] | 46.5 [26 to 68] | 49.5 [49 to 72] | 48.7 [37 to 57] | 48.1 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 17 | 16 | 6 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 4
  Not Hispanic or Latino | 16 | 13 | 6 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 11 | 6 | 29
  White | 2 | 1 | 0 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 6 | 39

OUTCOME MEASURES:

1. Primary Outcome: Collect Preliminary Data on In-vehicle Excess Particulate Matter (PM) Exposure
Description: monitor/report the PM levels as time-averaged sample (hourly averages) that will be monitored at work site and at homes across all groups
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Intervention Group | Wait-list Control Group | Peer Non-driver
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Group | Wait-list Control Group | Peer Non-driver
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/6
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT02381626/Prot_SAP_001.pdf